CLINICAL TRIAL: NCT06927713
Title: A Multi-center Randomised Controlled Trial to Explore the Ideal Stimulation Strategies at Hand Twelve Jing-Well Points in Patients With Disorders of Consciousness
Brief Title: Hand Jing-Well Points Stimulation to Treat Disorders of Consciousness
Acronym: Wells-DoC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY20252094JIANGWEN
Record Dates: First submitted 2025-03-30; First posted 2025-04-15 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-05

CONDITIONS: Disorders of Consciousness Due to Severe Brain Injury
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bloodletting Puncture (Experimental): Bloodletting puncture at hand twelve jing-well points for 5 consecutive days, once a day, combined with conventional medical treatment.
  Interventions: Other: Bloodletting Acupuncture
- Transcutaneous electrical stimulation (Experimental): Transcutaneous electrical acupoint stimulation at hand twelve jing-well points for 5 consecutive days, once a day, combined with conventional medical treatment.
  Interventions: Device: Transcutaneous electrical stimulation
- Control (No Intervention): Control group was treated with conventional medical treatment.

INTERVENTIONS:
Other: Bloodletting Acupuncture — Bloodletting was applied to the right hand ﬁrst and then the left hand in the order of Shaoshang (LU 11), Shangyang (LI 1), Zhongchong (PC 9), Guanchong (TE 1), Shaochong (HT 9) and Shaoze (SI 1).
  Arms: Bloodletting Puncture
Device: Transcutaneous electrical stimulation — Transcutaneous electrical acupoint stimulation at hand twelve jing-well points.
  Arms: Transcutaneous electrical stimulation

SUMMARY:
The purpose of this academic lead study is to explore the ideal stimulation strategies at Hand twelve jing-well points in patients with disorders of consciousness.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80 years old
* From 7 to 90 days since brain injury
* Diagnosed in VS/UWS or MCS as deﬁned by at least two CRS-R assessments performed during the screening period
* Acquired cerebral damage of known etiology
* Intact hand skin
* Informed consent given by the legal surrogate

Exclusion Criteria:

* Patients who continuously receive sedative drugs and Na+ or Ca2+ channel blockers (e.g., carbamazepine) or NMDA receptor antagonists (e.g., dextromethorphan)
* History of previous serious、progressive neurological disorder prior to the brian injury
* Epilepsy and seizure
* Unstable vital signs or life-threatening comorbidities
* Active implant (e.g., cardiac pacemakers/defibrillators, deep brain stimulators, ventriculoperitoneal shunt, etc)
* Documented pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised (CRS-R) change | baseline, immediately after the end of the 5-day treatment
  CRS-R score ranges from 0 to 23, with higher scores mean a better outcome.

SECONDARY OUTCOMES:
ABCD model change | baseline, immediately after the end of the 5-day treatment
  This model classifies the power spectrum of resting-state EEG data into four categories: A, B, C, and D. Type A exhibits a power spectrum peak in the delta range (0-4 Hz), indicative of a completely disconnected thalamocortical network. Type B shows a primary power spectrum peak in the theta range (4-8 Hz), reflecting a severely disconnected thalamocortical network. Type C exhibits power spectrum peaks in both the theta (4-8 Hz) and beta (13-24 Hz) ranges, indicative of a moderately disconnected thalamocortical network. Type D shows power spectrum peaks in the alpha (8-13 Hz) and beta ranges, representing a fully intact thalamocortical network.
ABCD model change | baseline, immediately after the end of the first treatment
  This model classifies the power spectrum of resting-state EEG data into four categories: A, B, C, and D. Type A exhibits a power spectrum peak in the delta range (0-4 Hz), indicative of a completely disconnected thalamocortical network. Type B shows a primary power spectrum peak in the theta range (4-8 Hz), reflecting a severely disconnected thalamocortical network. Type C exhibits power spectrum peaks in both the theta (4-8 Hz) and beta (13-24 Hz) ranges, indicative of a moderately disconnected thalamocortical network. Type D shows power spectrum peaks in the alpha (8-13 Hz) and beta ranges, representing a fully intact thalamocortical network.
Coma Recovery Scale-Revised (CRS-R) change | baseline, immediately after the end of the first treatment
  CRS-R score ranges from 0 to 23, with higher scores mean a better outcome.
Glasgow Outcome Scale-Extended (GOSE) | at six months post enrollment
  A GOSE score of 1 indicates death, 2 indicates a vegetative state, 3 to 4 indicates severe disability, 5 to 6 indicates moderate disability, and 7 to 8 indicates good recovery. Favorable functional outcome is deﬁned as an GOSE score of 4-8, while unfavorable functional outcome is defined as an GOSE score of 1-3.
Consciousness level change | baseline, at six months post enrollment
  The level of consciousness was evaluated using CRS-R score. Patients who transitioned from UWS to MCS (UWS-MCS) or to emergence from MCS (EMCS) (UWS-EMCS), from MCS minus to MCS plus (MCS - -MCS + ) or to EMCS (MCS - -EMCS), and from MCS to EMCS (MCS-EMCS) were categorized in the improved consciousness group. The unimproved consciousness was defined as a reduced or unchanged level of consciousness.
Correlation between EEG responsiveness and long-term outcomes | on the first day, the fifth day and at six months post enrollment
  EEG responsiveness to the treatment was considered positive if, after the hand Jing-Well points stimulation, patients exhibited elevated levels of EEG "ABCD" patterns compared to the baseline after either the first or fifth stimulation session. The correlation between EEG responsiveness and long-term consciousness improvement and favorable functional outcome was assessed.
Incidence of Adverse Events | from the first treatment to the end of the fifth treatment
  The incidence of adverse events occurred during the intervention period, including treatment intolerance：painful facial expressions, moans, crying, and head movements；Local adverse effect：skin infections (redness, swelling, suppuration), subcutaneous ecchymosis, skin burns (blisters or eschar formation)；Systemic adverse effect：epileptic seizures。

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China